CLINICAL TRIAL: NCT02899754
Title: Incorporating Veterans Preferences Into Lung Cancer Screening Decisions
Brief Title: Incorporating Veterans' Preferences Into Lung Cancer Screening Decisions
Acronym: LCSDecTool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIR 15-143
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer Screening
Keywords: lung cancer; decision support; implementation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm will use the lung cancer screening decision aid (LCSDecTool)
  Interventions: Behavioral: Lung Cancer Screening Decision Tool
- Control Group (Active Comparator): Content that provides general information on disease prevention and health promotion unrelated to lung cancer. The information will be delivered on the same modality and take a similar amount of time to administer.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Lung Cancer Screening Decision Tool — This will be a lung cancer screening decision support tool that is web based and provides patients with information about the potential benefits and harms associated with lung cancer screening and helps them to consider their personal values when making a decision about whether to initiate or continue with lung cancer screening.
  Other Names: LCSDecTool
  Arms: Intervention Group
Behavioral: Control Intervention — This will be a health message regarding prevention and healthy behavior that is not related to lung cancer screening but delivered in a similar modality and taking approximately the same amount of time as the LCSDecTool.
  Other Names: Control
  Arms: Control Group

SUMMARY:
Veterans have a high risk of developing lung in comparison to general populations due to their older age and smoking history. Recent evidence indicates that lung cancer screening with low dose CT scan reduces lung cancer mortality among older heavy smokers. However, the rates of false positive findings are high, requiring further testing and evaluation. The aims of this study were to 1) elicit patient and provider stakeholder input to inform the development of a lung cancer screening decision tool, 2) develop a web-based Lung Cancer Screening Decision Tool (LCSDecTool) that incorporates patient and provider input, and 3) conduct a RCT to evaluate LCSDecTool compared to usual care knowledge about LCS, decisional conflict and uptake of LCS.

The investigators hypothesized that the use of the LCSDecTool would decrease decisional conflict at 1 month. As a secondary outcome the investigators hypothesized that there would be a decrease in uptake of LCS in the LCDDecTool group compared with the control intervention due to increased awareness of harms associated with LCS. Additional secondary outcomes were LCS knowledge, decisional regret, anxiety, and lung cancer worry.

Veterans who were receiving primary care in a participating VA Medical Center, aged 55 to 80 years with a smoking history of at least 30 pack-years who were current smokers or had quit within the past 15 years were eligible to participate in the study.

Participants were asked to link on to a study website and were randomly assigned to the LCSDecTool or a control intervention website. Following use of the intervention, participants had a primary care visit. Patient reported outcomes were assessed immediately post intervention and at 1 and 3-months post intervention. LCS uptake was assessed at 6 months post-intervention.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths in the United States. Recent clinical trials provide evidence that screening with low dose CT scans will decrease lung cancer and all-cause mortality among older heavy smokers. Clinical guidelines have been issued with the USPSTF recommending annual screening from age 55 to 80 for those with 30 pack years or more of smoking or who quit less than 15 years ago. Evidence clearly delineates both the benefits (mortality reduction) and harms (false positives, follow-up testing, risk of invasive testing, and risk of overdiagnosis) of lung cancer screening. Preliminary data from an HSR&D pilot grant finds that some Veterans are highly reluctant to enter the care pathway associated with lung cancer screening due to its potential harms. Additional preliminary data using Best Worst Scaling in older smokers demonstrate groups of patients who place greater importance on harms than benefit when considering lung cancer screening. Preference assessment methods can help Veterans to weigh benefits and harms, consider the clinical pathway they are entering, anticipate future health states, and communicate these values to their health care providers. Although basic educational tools to inform lung cancer decision-making have been developed, there is a lack of validated preference assessment tools that can be integrated into the clinical setting. Building upon preference assessment methods developed and validated in an HSR&D pilot grant (PI-Schapira) and using a trans-disciplinary approach, this team is positioned to advance the science and practice of decision support for lung cancer screening in the Veteran population. The objectives of this study are to 1) elicit patient and provider stakeholder input to inform the development of a lung cancer screening decision tool, 2) develop a web based Lung Cancer Screening Decision Tool (LCSDecTool) that incorporates patient and provider input, and 3) evaluate the impact of the LCSDecTool compared to usual care on the decision process, clinical outcomes, and quality of life. The study will be conducted in 3 phases. In phase 1, mixed methods will be used to assess usability of preference assessment methods and perceived usefulness of a web based lung cancer screening decision support tool among patient and provider stakeholders. In phase 2, an interactive web based decision support program will be developed that incorporates preference assessment methods. In phase 3, a pilot RCT will be conduced to evaluate the efficacy of the web based decision support program. Outcomes evaluated will include decision quality as indicated by knowledge, decisional conflict, and decision regret; screening behavior, clinical outcomes as indicated by anxiety, and quality of life. The study was conducted across three VA sites; West Haven-VA in Connecticut, Corporal Michael J. Crescenz VA in Philadelphia, Pennsylvania, and the Zablocki VA in Milwaukee, WI. Results of this study will provide tools that can be used to integrate lung cancer screening into clinical practice at VA Medical Centers in a patient centered approach. Lung cancer screening is fundamentally different from existing screening paradigms in several respects; eligibility is defined by a behavior (smoking), a high rate of false positive findings is expected, and the target population is older with higher comorbidity than the target population for cervical, breast, or colorectal screening. Given these unique aspects of lung cancer screening, there is a critical need to develop and test tools for preference assessment and informed decision making that are applicable for the VA setting. The current proposal provides a mechanism to accomplish these goals. The Principal Investigator is working closely with the US Department of Veterans Affairs National Center for Health Promotion and Disease Prevention to integrate the tools and paradigm developed to primary care in the VA Medical Care System. The work builds directly upon a recently completed HSR&D pilot support in the area of lung cancer and shared decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80 years
* Enrolled in a Patient Aligned Care Team at a participating site
* 30 or more pack years of smoking
* Active smoker or quit smoking within 15 years

Exclusion Criteria:

* Cognitive impairment as determined by clinical history
* Previous diagnosis of cancer with the exception of non-melanoma skin cancer and localized prostate cancer that is 1-year post-diagnosis
* Life expectancy of less than 2 years as indicated by chart review and conformation with PCPC
* Inability to speak English
* Active surveillance of Lung Nodule,
* Enrolled in CMCVAMC Lung Cancer Screening Program

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn M. Schapira, MD MPH, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA; Jeffrey C Whittle, MD MPH, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (3):
- United States (3):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) that indicates adherence to any applicable Informed Consent provisions, appropriately limits use of the dataset and prohibits the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
  A De-identified, Anonymized Dataset will be created and shared.
  A limited coded dataset will be made available on our CMCVAMC research website that is publically available.
  The dataset will be housed on a server, administered by CHERP behind the VA firewall, access being granted only to those who apply directly to the principal investigator , provide the necessary assurances that they will not re-identify the data, and submit to a clearance by the CMCVAMC Privacy Officer

REFERENCES:
- [Background] Schapira MM. The Conundrum and Challenge of Lung Cancer Screening Shared Decision-making Implementation. J Gen Intern Med. 2018 Jul;33(7):989-990. doi: 10.1007/s11606-018-4449-z. No abstract available. PMID 29736754
- [Background] Kim RY, Rendle KA, Mitra N, Saia CA, Neslund-Dudas C, Greenlee RT, Burnett-Hartman AN, Honda SA, Simoff MJ, Schapira MM, Croswell JM, Meza R, Ritzwoller DP, Vachani A. Racial Disparities in Adherence to Annual Lung Cancer Screening and Recommended Follow-Up Care: A Multicenter Cohort Study. Ann Am Thorac Soc. 2022 Sep;19(9):1561-1569. doi: 10.1513/AnnalsATS.202111-1253OC. PMID 35167781
- [Background] Schapira MM, Rendle KA. Rising to the De-escalation Challenge: Multilevel Change Needed to Align Clinical Practice with Cancer Screening Guidelines. Med Decis Making. 2022 Nov;42(8):1045-1047. doi: 10.1177/0272989X221125168. No abstract available. PMID 36255190
- [Result] Schapira MM, Rodriguez KL, Chhatre S, Fraenkel L, Bastian LA, Kravetz JD, Asan O, Akers S, Vachani A, Prigge JM, Meline J, Ibarra JV, Corn B, Kaminstein D. When Is a Harm a Harm? Discordance between Patient and Medical Experts' Evaluation of Lung Cancer Screening Attributes. Med Decis Making. 2021 Apr;41(3):317-328. doi: 10.1177/0272989X20987221. Epub 2021 Feb 6. PMID 33554740
- [Result] Schapira MM, Hubbard RA, Whittle J, Vachani A, Kaminstein D, Chhatre S, Rodriguez KL, Bastian LA, Kravetz JD, Asan O, Prigge JM, Meline J, Schrand S, Ibarra JV, Dye DA, Rieder JB, Frempong JO, Fraenkel L. Lung Cancer Screening Decision Aid Designed for a Primary Care Setting: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2330452. doi: 10.1001/jamanetworkopen.2023.30452. PMID 37647070
- See also: This website hosts lung cancer screening educational materials developed by the VA that will be used in the study — http://www.prevention.va.gov/preventing_diseases/screening_for_lung_cancer.asp

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 69 | 71
Completed | 62 (Our primary outcome was at T2 where we had 62 completed) | 62 (Our primary outcome was at t2 where we had 62 completed)
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [61.0 to 69.0] | 65.0 [62.0 to 70.0] | 64.0 [61.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 61 | 68 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 68 | 68 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 33 | 75
  White | 26 | 36 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 71 | 140
Education [Count of Participants; unit: Participants]
  Grade School | 3 | 1 | 4
  High School | 28 | 24 | 52
  Some College or University | 33 | 39 | 72
  Four or more years of college or university | 3 | 6 | 9
  Post-college graduate degree | 2 | 1 | 3
Income [Count of Participants; unit: Participants]
  0-25,000 | 28 | 15 | 43
  >25,000 - 50.000 | 24 | 32 | 56
  >50.000 - 75,000 | 11 | 9 | 20
  >75.000 - 100.000 | 1 | 3 | 4
  >100.000 | 2 | 3 | 5
  Prefer not to say | 3 | 9 | 12
Post Traumatic Stress Syndrome [Count of Participants; unit: Participants]
  Post-Traumatic Stress Syndrome Yes | 31 | 31 | 62
  Post-Traumatic Stress Syndrome No | 38 | 40 | 78
Depression [Count of Participants; unit: Participants]
  Depression Yes | 33 | 28 | 61
  Depression No | 36 | 43 | 79
Anxiety [Count of Participants; unit: Participants]
  Anxiety Yes | 24 | 23 | 47
  Anxiety No | 45 | 48 | 93
Hypertension [Count of Participants; unit: Participants]
  Hypertension Yes | 25 | 24 | 49
  Hypertension No | 44 | 47 | 91
Diabetes [Count of Participants; unit: Participants]
  Diabetes Yes | 18 | 23 | 41
  Diabetes No | 51 | 48 | 99
Emphysema [Count of Participants; unit: Participants]
  Emphysema Yes | 14 | 14 | 28
  Emphysema No | 55 | 57 | 112
Heart Disease [Count of Participants; unit: Participants]
  Heart Disease Yes | 9 | 17 | 26
  Heart Disease No | 60 | 54 | 114
Asthma [Count of Participants; unit: Participants]
  Asthma Yes | 4 | 3 | 7
  Asthma No | 65 | 68 | 133
Health Literacy [Median (Inter-Quartile Range); unit: units on a scale] — Baseline measures included health literacy assessed by the Rapid Estimate of Adult Literacy in Medicine scale which asks respondents to read and pronounce 66 medically related words, is scored from 0 to 66 (higher scores indicate greater health literacy) and categorizes persons in terms of grade level reading skills.
  Below are the range of scores that correlate to reading grade level.
  Score: 0-18 (≤3rd grade) Score 19-44 (4th-5th grade) Score 45-60 (6th-7th grade) Score 61-66 (8th-9th grade)
  units on a scale | 66.0 [66.0 to 66.0] | 66.0 [65.0 to 66.0] | 66.0 [65.0 to 66.0]
Numeracy [Median (Inter-Quartile Range); unit: units on a scale] — Health numeracy was assessed with the Numeracy Understanding in Medicine Instrument Short Form, an 8-item scale with scores ranging from 0 (low numeracy) to 8(high numeracy).
  units on a scale | 4.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
Arthritis [Count of Participants; unit: Participants]
  Arthritis Yes | 30 | 35 | 65
  Arthritis No | 39 | 36 | 75
Smoking Pack Years [Median (Inter-Quartile Range); unit: Pack Years of Smoking] | 40.8 [35.0 to 50.0] | 46.0 [39.5 to 54.2] | 44.2 [37.5 to 52.0]

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict
Description: The Decisional Conflict Scale is a 16-item scale with a value that ranges 0 (low decisional conflict) to 100 (high decisional conflict. The scale includes five subscales in the domains of uncertainty ( 3 items), Informed (3 items), Value Clarity (3 items), Support ( 3 items), and Effective DM (4 items).
  Each item is scored from a 0 (strongly agree), 1 (agree), 2 (neither agree nor disagree), 3) (disagree) or 4 (strongly disagree). The total sore for the 16 items is calculated by a) summing scores, b) dividing by 16, c) multiplying by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
  For each subscale the scores are obtained by a) summing scores, b) dividing by the number of items in the subscale, c) multiplying by 25. Scores are interpreted as range from 0(low decisional conflict) to 100 (high decisional conflict) in the respective domains.
Time Frame: 1 month following the intervention
Population: There were 7 participants that were lost to follow-up at the 1 month visit in the experimental group and 9 participants that were lost to follow up at the 1 month visit in the control group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 62 | 62
units on a scale | 25.7 [21.4 to 30.1] | 29.9 [25.6 to 34.2]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Primary outcome assessed at 1 month post-intervention; Test type: Superiority; p = 0.18, t-test, 2 sided

2. Secondary Outcome: Decision Regret
Description: Decision regret as measured by a 5-item Decision Regret scale that is patient reported. This score range is from 0 (low decisional regret) to 100 (high decisional regret).
Time Frame: 1 month following intervention
Population: There were 7 participants that were lost to follow-up at the 1 month follow-up visit in experimental intervention group and 9 participants in the control group that were lost to follow up at the 1 month follow-up visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 62 | 62
units on a scale | 34.7 [32.2 to 37.2] | 32.2 [29.6 to 34.8]

3. Secondary Outcome: Lung Cancer Knowledge
Description: Knowledge was measured with the 12-Item Brief Measures of Smokers Knowledge of Lung Cancer Screening Scale. The scores on this scale range from 0 (low level of knowledge) to 12 (high level of knowledge). Higher scores indicate a better outcome. Each correct response to an item is added to create the final score.
Time Frame: Immediately Post Intervention, within 24 hours of intervention following the intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 69 | 71
units on a scale | 7.0 [6.3 to 7.7] | 4.9 [4.3 to 5.5]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p < 0.01, t-test, 2 sided

4. Secondary Outcome: Lung Cancer Screening Knowledge
Description: Knowledge was measured with the 12-Item Brief Measures of Smokers Knowledge of Lung Cancer Screening Scale. The scores on this scale range from 0 (low level of knowledge) to 12 (high level of knowledge). Higher scores indicate a higher amount of knowledge. Higher scores are a better outcome. 1 point is given to each correct item. The points are added to provide the total score.
Time Frame: 1 month post intervention
Population: There were 7 participants that were lost to follow up at the time of the 1 month survey assessment for the experimental group and 9 participants lost to follow-up at the time of the 1 month survey assessment.in the control group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 62 | 62
units on a scale | 6.3 [5.7 to 6.8] | 5.2 [4.5 to 5.8]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.02, t-test, 2 sided

5. Secondary Outcome: Lung Cancer Screening Knowledge
Description: Knowledge was measured with the 12-Item Brief Measures of Smokers Knowledge of Lung Cancer Screening Scale. The scores on this scale range from 0 (low level of knowledge) to 12 (high level of knowledge).
Time Frame: 3 months post intervention
Population: There were 9 participants in the experimental group that were lost to follow-up at the time of the 3 month survey and 14 participants in the control group that were lost to follow-up at the time of the 3 month survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 60 | 57
units on a scale | 6.2 [5.6 to 6.8] | 5.1 [4.4 to 5.8]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.01, t-test, 2 sided

6. Secondary Outcome: Anxiety
Description: State anxiety was measured on the State Trait Anxiety Index Scale using the State subscale. This measure included 20 items with a total score ranging from 20 (low anxiety) to 80 (high anxiety).
Time Frame: 1 month following intervention
Population: There were 7 participants in the experimental intervention group that were lost to follow up at the 1 month survey assessment and 9 participants in the control group that were lost to follow up at the 2 month survey assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 62 | 62
units on a scale | 37.2 [34.0 to 40.4] | 35.2 [31.3 to 39.0]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.22, t-test, 2 sided

7. Secondary Outcome: Lung Cancer Screening Uptake
Description: Documentation of receiving a lung cancer screening test by 6 months following the intervention. This was obtained by chart review.
Time Frame: 6 months after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 69 | 71
Participants | 26 | 15
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.18, t-test, 2 sided

8. Secondary Outcome: Lung Cancer Screening Uptake Within 9 Months
Description: A documented lung cancer screening test completed within 9 months of the intervention obtained by chart review
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 69 | 71
Participants | 31 | 18
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; chi-square test; Test type: Superiority; p = 0.01, Chi-squared

9. Secondary Outcome: Lung Cancer Worry
Description: Lung cancer worry as measured by a 7 item scale with a range of scores from 3 (low worry) to 13 (high worry).
Time Frame: 1 month after the intervention
Population: There were 7 participants in the experimental intervention group that were lost to follow-up at the 1 month survey and 9 participants in the control group that were lost to follow-up at the 1 month survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 62 | 62
units on a scale | 6.3 [5.7 to 6.8] | 6.3 [5.7 to 7.0]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.64, t-test, 2 sided

10. Secondary Outcome: Decisional Conflict
Description: Measured by the Decisional Conflict Scale a 16-item scale with scores from 0(low decisional conflict) to 100 (high decisional conflict).
Time Frame: Immediately post-intervention-the same day as the intervention following the intervention.
Population: Two participants in the intervention group did not complete the immediately post-intervention survey and 2 participants in the control group did not complete the immediately post-intervention survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 69
units on a scale | 22.2 [18.3 to 26.0] | 31.1 [26.1 to 36.0]

11. Secondary Outcome: Decisional Conflict
Description: Decisional conflict as measured by the 16 item decisional conflict scale scored from 0 (low decisional conflict) to 100 (high decisional conflict)
Time Frame: 3 months post-intervention
Population: There were 9 participants that were lost to follow-up at the 3 month survey assessment in the intervention group and 14 lost to follow-up at the 3 month assessment in the control group.
Measure: Mean (95% Confidence Interval); unit: Scores on the decisional conflict scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 60 | 57
Scores on the decisional conflict scale | 24.2 [20.8 to 27.6] | 27.5 [23.3 to 31.7]

12. Secondary Outcome: Decisional Regret
Description: Decisional regret was measured on the Decisional Regret scale. This is a 5 time scale with scores ranging from 0 (low decisional regret) to 100 (high decisional regret).
Time Frame: 3 months post-intervention
Population: There were 9 participants lost to follow-up from the intervention group at the 3 month survey and 14 participants lost to follow-up in the intervention group at the 3 month survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 60 | 57
units on a scale | 32.5 [30.1 to 35.0] | 34.3 [31.9 to 36.7]

13. Secondary Outcome: Decisional Regret
Description: Decisional regret was measured on a 5 point decisional regret scale with scores ranging from 0 (low regret) to 100 (high regret).
Time Frame: Immediately post-intervention-the same day as the intervention following the intervention
Population: There were 2 participants in the intervention group and 2 participants in the control group that did not complete the post-intervention survey when this outcome was ascertained.
Measure: Mean (95% Confidence Interval); unit: Score on Decisional Regret Scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 69
Score on Decisional Regret Scale | 32.6 [30.1 to 35.1] | 34.5 [31.9 to 37.1]

14. Secondary Outcome: Anxiety
Description: Trait anxiety was measured using the State Trait Anxiety Index. This is a 20 item measure with scores ranging from 20 (low anxiety) to 80 (high anxiety).
Time Frame: Immediately post-intervention-the same day as the intervention following the intervention
Population: There were 2 participants in the intervention group that did not complete the immediately post intervention survey and 2 participants in the control group that did not complete the immediately post-intervention survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 69
units on a scale | 33.5 [30.7 to 36.3] | 32.8 [29.8 to 35.9]

15. Secondary Outcome: Anxiety
Description: Anxiety was measured using the Trait items on the State Trait Anxiety Index with scores ranging from 20 (low anxiety) to 80 (high anxiety).
Time Frame: 3 months post intervention
Population: There were 9 participants in the intervention group that did not complete the 3 months follow up survey and 14 participants in the control group that did not complete the 3 months follow-up survey.
Measure: Mean (95% Confidence Interval); unit: Scores on the State Trait Anxiety Index
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 60 | 57
Scores on the State Trait Anxiety Index | 36.6 [33.6 to 39.7] | 38.2 [33.9 to 42.4]

16. Secondary Outcome: Lung Cancer Worry
Description: Lung cancer worry was measured on a 3 point scale with scores ranging from 3 (low worry) to 13 (high worry)
Time Frame: immediately post-intervention-the same day as the intervention following the intervention.
Population: There were 2 participants in the intervention group and 2 participants in the control group that did not complete the immediately post-intervention survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 69
units on a scale | 5.9 [5.2 to 6.5] | 6.4 [5.9 to 6.9]

17. Secondary Outcome: Lung Cancer Worry
Description: Lung Cancer Worry was measured on a 3 item scale with scores ranging from 3(low worry) to 13 (high worry)
Time Frame: 3 months post-intervention
Population: There were 9 participants in the intervention group and 14 participants in the control group that did not complete the 3 months post-intervention survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 60 | 57
units on a scale | 5.4 [4.9 to 6.0] | 5.9 [5.3 to 6.6]

ADVERSE EVENTS:
Time Frame: The investigators monitored for adverse events from the date each patient was enrolled to 9 months following the completion of the each patients' intervention visit.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/71
Other Adverse Events (participants affected / at risk) | 0/69 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT02899754/Prot_SAP_000.pdf
  • Informed Consent Form: Oral Consent Form Option (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02899754/ICF_001.pdf
  • Informed Consent Form: Written Consent Form Option (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02899754/ICF_002.pdf